CLINICAL TRIAL: NCT04397211
Title: Comparison of Angiography-derived Fractional FLow Reserve- And IntraVascular Ultrasound-guided Intervention Strategy for Clinical OUtcomes in Patients With CoRonary Artery Disease
Brief Title: Angiography-Derived FFR And IVUS for Clinical Outcomes in Patients With Coronary Artery Disease
Acronym: FLAVOUR II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Seoul National University Hospital (Other); Affiliated Hangzhou First People's Hospital (Unknown); Wuhan University (Other); Peking University Third Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); RenJi Hospital (Other); Second Hospital of Shanxi Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Changxing People's Hospital (Other); The Affiliated Hospital of Medical College, Ningbo University (Other); Jinhua Central Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Dongyang People's Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Jining First People's Hospital (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Ulsan University Hospital (Other); Huizhou Municipal Central Hospital (Other); Zhejiang Greentown Cardiovascular Hospital (Other); The Fourth People's Hospital of Jinan (Unknown); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-303
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: Angiography-derived fractional flow reserve; Intravascular ultrasound; Percutaneous coronary intervention; Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography-derived FFR-guided PCI group (Active Comparator): Percutaneous coronary intervention using drug-eluting stent(s) will be performed by Angiography-derived FFR-guided strategy
  Interventions: Procedure: Angiography-derived FFR
- IVUS-guided PCI group (Active Comparator): Percutaneous coronary intervention using drug-eluting stent(s) will be performed by IVUS-guided strategy
  Interventions: Procedure: IVUS

INTERVENTIONS:
Procedure: Angiography-derived FFR — The percutaneous coronary intervention using drug-eluting stent will be indicated according to following criteria in the Angiography-derived FFR-guided strategy arm
  *Criteria for revascularization: Angiography-derived FFR ≤ 0.80
  Arms: Angiography-derived FFR-guided PCI group
Procedure: IVUS — The percutaneous coronary intervention using drug-eluting stent will be indicated according to following criteria in the IVUS-guided strategy arm
  *Criteria for revascularization: Minimum lumen area (MLA) ≤ 3mm2 or 3< MLA ≤ 4mm2 & Plaque burden > 70%
  Arms: IVUS-guided PCI group

SUMMARY:
Comparison of Angiography-derived Fractional FLow Reserve And IntraVascular Ultrasound-guided Intervention Strategy for Clinical OUtcomes in Patients with CoRonary Artery Disease

DETAILED DESCRIPTION:
1. The primary hypothesis is that angiography-derived FFR-guided strategy for PCI with a drug-eluting stent (DES) will show non-inferiority in rates of patients-oriented composite outcomes (POCO) at 12 months after randomization, compared with IVUS-guided strategy for PCI with a DES in patients with coronary artery disease.
2. Study population and sample size calculation： Sample size calculation based on the event rates of previous trials, investigators predicted the rates of POCO at 12 months after PCI will be 7% in the Angiography-derived FFR-guided arm, and 8% in the IVUS-guided arm

   * Primary endpoint: patient-oriented composite outcome (a composite of all-cause death, MI, any revascularization) at 12 months after PCI
   * Design: non-inferiority, delta = 2.5%
   * Sampling ratio: angiography-derived FFR-guided strategy: IVUS-guided strategy = 1:1
   * Type I error (α): One-sided 2.5%
   * Accrual time: 3 years
   * Total time: 4 years (accrual 3 years + follow-up 1 years)
   * Assumption: POCO 7.0% vs. 8.0% in angiography-derived FFR or IVUS-guided strategy, respectively
   * Statistical power (1- β): 80%
   * Primary statistical method: Kaplan-Meier survival analysis with log-rank test
   * Estimated attrition rate: total 5%
   * Stratification in Randomization: Presence of diabetes mellitus (35% of patients in each group) Based on the above assumption, we would need total 1,872 patients (936 patients in each group) with consideration of an attrition rate.
3. Research Materials and Indication for Revascularization： For the angiography-derived FFR-guided strategy arm, criteria for revascularization: angiography-derived FFR ≤ 0.80. For the IVUS-guided strategy arm, the criterion for revascularization is MLA ≤ 3mm2 or [3mm2 < MLA ≤ 4mm2 and plaque burden > 70%].

ELIGIBILITY:
Inclusion Criteria:

* ① Subject must be ≥ 18 years. ② Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and PCI with a drug-eluting stent (DES) and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure. ③ Patients suspected with ischemic heart disease. ④ Patients with ≥ 50% stenosis by angiography-based visual estimation eligible for stent implantation. ⑤ Target vessel size ≥ 2.5mm in visual estimation. ⑥ Target vessels are limited to major epicardial coronary arteries (left anterior descending artery[LAD], left circumflex artery [LCX], right coronary artery [RCA])

Exclusion Criteria:

* ① The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled.) ② Patients with active pathologic bleeding. ③ Gastrointestinal or genitourinary major bleeding within the prior 3 months. ④ History of bleeding. diathesis, known coagulopathy (including heparin-induced thrombocytopenia). ⑤Non-cardiac co-morbid conditions with life expectancy < 1 year. ⑥ Target vessel total occlusion. ⑦ Target lesion located in coronary arterial bypass graft. ⑧ Left main coronary artery stenosis ≥ 50%. ⑨ Not eligible for angiography-derived FFR (ostial RCA ≥ 50% stenosis, myocardial bridging, severe tortuosity, severe overlap, poor image quality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1872 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | 12 months
  Patient-oriented composite outcome (POCO), defined as a composite of all death, myocardial infarction (MI) or any revascularization at 12 months after randomization according to the ARC definitions.

SECONDARY OUTCOMES:
Patient-oriented composite outcome (POCO) | 24, 60 months
  POCO at 24 and 60 months after randomization according to the ARC consensus
Target vessel failure | 12, 24 and 60 months
  Target vessel failure (a composite of cardiac death, target-vessel MI, or target vessel revascularization)
Cost-effectiveness analysis | 12, 24 and 60 months
  Cost-effectiveness analysis
All-cause and cardiac death | 12, 24 and 60 months
  All-cause and cardiac death
Any nonfatal MI without peri-procedural MI | 12, 24 and 60 months
  Any nonfatal MI without peri-procedural MI
Any nonfatal MI with peri-procedural MI | 12, 24 and 60 months
  Any nonfatal MI with peri-procedural MI
Any target vessel/lesion revascularization | 12, 24 and 60 months
  Any target vessel/lesion revascularization
Any non-target vessel/lesion revascularization | 12, 24 and 60 months
  Any non-target vessel/lesion revascularization
Any revascularization (ischemia-driven or all) | 12, 24 and 60 months
  Any revascularization (ischemia-driven or all)
Stent thrombosis (definite/probable/possible) | 12, 24 and 60 months
  Stent thrombosis (definite/probable/possible)
Stroke (ischemic and hemorrhagic) | 12, 24 and 60 months
  Stroke (ischemic and hemorrhagic)
Acute success of procedure and rate of PCI optimization | At discharge (1 week after index procedure)
  Acute success of procedure and rate of PCI optimization

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (23):
- China (21):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - Second Affiliated Hospital of Shantou University Medical College, Guangdong
  - Affiliated Hangzhou First People's Hospital, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou
  - Changxing People's Hospital, Huzhou
  - Huzhou Central Hospital, Huzhou
  - The Fourth People's Hospital of Jinan, Jinan
  - Dongyang People's Hospital, Jinhua
  - Jinhua Central Hospital, Jinhua
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Hospital of Medical College, Ningbo University, Ningbo
  - Shandong Jining No.1 People's Hospital, Shandong
  - Shandong University of Traditional Chinese Medicine, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Second hospital of Shanxi Medical University, Taiyuan
  - The first affiliated hospital of Wenzhou Medical University, Wenzhou
  - The second affiliated hospital of Wenzhou Medical University, Wenzhou
  - Zhongnan Hospital of Wuhan University, Wuhan
- South Korea (2):
  - Seoul National University Hospital,, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Result] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Result] Melikian N, De Bondt P, Tonino P, De Winter O, Wyffels E, Bartunek J, Heyndrickx GR, Fearon WF, Pijls NH, Wijns W, De Bruyne B. Fractional flow reserve and myocardial perfusion imaging in patients with angiographic multivessel coronary artery disease. JACC Cardiovasc Interv. 2010 Mar;3(3):307-14. doi: 10.1016/j.jcin.2009.12.010. PMID 20298990
- [Result] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Result] Westra J, Tu S, Campo G, Qiao S, Matsuo H, Qu X, Koltowski L, Chang Y, Liu T, Yang J, Andersen BK, Eftekhari A, Christiansen EH, Escaned J, Wijns W, Xu B, Holm NR. Diagnostic performance of quantitative flow ratio in prospectively enrolled patients: An individual patient-data meta-analysis. Catheter Cardiovasc Interv. 2019 Nov 1;94(5):693-701. doi: 10.1002/ccd.28283. Epub 2019 Apr 9. PMID 30963676
- [Result] Fearon WF, Achenbach S, Engstrom T, Assali A, Shlofmitz R, Jeremias A, Fournier S, Kirtane AJ, Kornowski R, Greenberg G, Jubeh R, Kolansky DM, McAndrew T, Dressler O, Maehara A, Matsumura M, Leon MB, De Bruyne B; FAST-FFR Study Investigators. Accuracy of Fractional Flow Reserve Derived From Coronary Angiography. Circulation. 2019 Jan 22;139(4):477-484. doi: 10.1161/CIRCULATIONAHA.118.037350. PMID 30586699
- [Result] Westra J, Tu S, Winther S, Nissen L, Vestergaard MB, Andersen BK, Holck EN, Fox Maule C, Johansen JK, Andreasen LN, Simonsen JK, Zhang Y, Kristensen SD, Maeng M, Kaltoft A, Terkelsen CJ, Krusell LR, Jakobsen L, Reiber JHC, Lassen JF, Bottcher M, Botker HE, Christiansen EH, Holm NR. Evaluation of Coronary Artery Stenosis by Quantitative Flow Ratio During Invasive Coronary Angiography: The WIFI II Study (Wire-Free Functional Imaging II). Circ Cardiovasc Imaging. 2018 Mar;11(3):e007107. doi: 10.1161/CIRCIMAGING.117.007107. PMID 29555835
- [Result] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Result] Collet C, Onuma Y, Sonck J, Asano T, Vandeloo B, Kornowski R, Tu S, Westra J, Holm NR, Xu B, de Winter RJ, Tijssen JG, Miyazaki Y, Katagiri Y, Tenekecioglu E, Modolo R, Chichareon P, Cosyns B, Schoors D, Roosens B, Lochy S, Argacha JF, van Rosendael A, Bax J, Reiber JHC, Escaned J, De Bruyne B, Wijns W, Serruys PW. Diagnostic performance of angiography-derived fractional flow reserve: a systematic review and Bayesian meta-analysis. Eur Heart J. 2018 Sep 14;39(35):3314-3321. doi: 10.1093/eurheartj/ehy445. PMID 30137305
- [Result] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Result] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Result] Fujii K, Carlier SG, Mintz GS, Yang YM, Moussa I, Weisz G, Dangas G, Mehran R, Lansky AJ, Kreps EM, Collins M, Stone GW, Moses JW, Leon MB. Stent underexpansion and residual reference segment stenosis are related to stent thrombosis after sirolimus-eluting stent implantation: an intravascular ultrasound study. J Am Coll Cardiol. 2005 Apr 5;45(7):995-8. doi: 10.1016/j.jacc.2004.12.066. PMID 15808753
- [Result] Ahn JM, Kang SJ, Yoon SH, Park HW, Kang SM, Lee JY, Lee SW, Kim YH, Lee CW, Park SW, Mintz GS, Park SJ. Meta-analysis of outcomes after intravascular ultrasound-guided versus angiography-guided drug-eluting stent implantation in 26,503 patients enrolled in three randomized trials and 14 observational studies. Am J Cardiol. 2014 Apr 15;113(8):1338-47. doi: 10.1016/j.amjcard.2013.12.043. Epub 2014 Jan 31. PMID 24685326
- [Result] Nam CW, Yoon HJ, Cho YK, Park HS, Kim H, Hur SH, Kim YN, Chung IS, Koo BK, Tahk SJ, Fearon WF, Kim KB. Outcomes of percutaneous coronary intervention in intermediate coronary artery disease: fractional flow reserve-guided versus intravascular ultrasound-guided. JACC Cardiovasc Interv. 2010 Aug;3(8):812-7. doi: 10.1016/j.jcin.2010.04.016. PMID 20723852
- [Result] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Result] Zhang J, Gao X, Kan J, Ge Z, Han L, Lu S, Tian N, Lin S, Lu Q, Wu X, Li Q, Liu Z, Chen Y, Qian X, Wang J, Chai D, Chen C, Li X, Gogas BD, Pan T, Shan S, Ye F, Chen SL. Intravascular Ultrasound Versus Angiography-Guided Drug-Eluting Stent Implantation: The ULTIMATE Trial. J Am Coll Cardiol. 2018 Dec 18;72(24):3126-3137. doi: 10.1016/j.jacc.2018.09.013. Epub 2018 Sep 24. PMID 30261237
- [Result] Park KW, Kang SH, Yang HM, Lee HY, Kang HJ, Cho YS, Youn TJ, Koo BK, Chae IH, Kim HS. Impact of intravascular ultrasound guidance in routine percutaneous coronary intervention for conventional lesions: data from the EXCELLENT trial. Int J Cardiol. 2013 Aug 10;167(3):721-6. doi: 10.1016/j.ijcard.2012.03.059. Epub 2012 Apr 4. PMID 22481046
- [Result] Kang J, Koo BK, Hu X, Lee JM, Hahn JY, Yang HM, Shin ES, Nam CW, Doh JH, Lee BK, Ahn C, Wang J, Tahk SJ. Comparison of Fractional FLow Reserve And Intravascular ultrasound-guided Intervention Strategy for Clinical OUtcomes in Patients with InteRmediate Stenosis (FLAVOUR): Rationale and design of a randomized clinical trial. Am Heart J. 2018 May;199:7-12. doi: 10.1016/j.ahj.2017.11.001. Epub 2017 Nov 6. PMID 29754669
- [Result] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Result] ISCHEMIA Trial Research Group; Maron DJ, Hochman JS, O'Brien SM, Reynolds HR, Boden WE, Stone GW, Bangalore S, Spertus JA, Mark DB, Alexander KP, Shaw L, Berger JS, Ferguson TB Jr, Williams DO, Harrington RA, Rosenberg Y. International Study of Comparative Health Effectiveness with Medical and Invasive Approaches (ISCHEMIA) trial: Rationale and design. Am Heart J. 2018 Jul;201:124-135. doi: 10.1016/j.ahj.2018.04.011. Epub 2018 Apr 21. PMID 29778671
- [Result] Maron DJ, Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Boden WE, Chaitman BR, Senior R, Lopez-Sendon J, Alexander KP, Lopes RD, Shaw LJ, Berger JS, Newman JD, Sidhu MS, Goodman SG, Ruzyllo W, Gosselin G, Maggioni AP, White HD, Bhargava B, Min JK, Mancini GBJ, Berman DS, Picard MH, Kwong RY, Ali ZA, Mark DB, Spertus JA, Krishnan MN, Elghamaz A, Moorthy N, Hueb WA, Demkow M, Mavromatis K, Bockeria O, Peteiro J, Miller TD, Szwed H, Doerr R, Keltai M, Selvanayagam JB, Steg PG, Held C, Kohsaka S, Mavromichalis S, Kirby R, Jeffries NO, Harrell FE Jr, Rockhold FW, Broderick S, Ferguson TB Jr, Williams DO, Harrington RA, Stone GW, Rosenberg Y; ISCHEMIA Research Group. Initial Invasive or Conservative Strategy for Stable Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1395-1407. doi: 10.1056/NEJMoa1915922. Epub 2020 Mar 30. PMID 32227755
- [Derived] Hu X, Zhang J, Yang S, Jiang J, Peng X, Lu D, Pan Y, Guo L, Li J, He W, Zhou H, Pu J, Huang J, Jiang F, Liu Q, Song D, Lu L, Cheng Z, Yang B, Ma J, Chen P, Li S, Meng Z, Tang L, Fan Y, Shin ES, Tu S, Nam CW, Fearon WF, Koo BK, Wang J; FLAVOUR II study group. Angiography-derived fractional flow reserve versus intravascular ultrasound to guide percutaneous coronary intervention in patients with coronary artery disease (FLAVOUR II): a multicentre, randomised, non-inferiority trial. Lancet. 2025 Apr 26;405(10488):1491-1504. doi: 10.1016/S0140-6736(25)00504-5. Epub 2025 Mar 30. PMID 40174597
- [Derived] Zhang J, Hu X, Jiang J, Lu D, Guo L, Peng X, Pan Y, He W, Li J, Zhou H, Huang J, Jiang F, Pu J, Cheng Z, Yang B, Ma J, Chen P, Liu Q, Song D, Lu L, Li S, Fan Y, Meng Z, Tang L, Shin ES, Tu S, Koo BK, Wang J. Rationale and design of a comparison of angiography-derived fractional flow reserve-guided and intravascular ultrasound-guided intervention strategy for clinical outcomes in patients with coronary artery disease: a randomised controlled trial (FLAVOUR II). BMJ Open. 2023 Dec 10;13(12):e074349. doi: 10.1136/bmjopen-2023-074349. PMID 38072492